CLINICAL TRIAL: NCT02201966
Title: Regional Interdependence of the Shoulders and Hips in Gymnasts With Low Back Pain
Status: Withdrawn | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mitchell Selhorst, Principle Investigator, Nationwide Children's Hospital
Other Study IDs: IRB14-00229
Record Dates: First submitted 2014-07-23; First posted 2014-07-28 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Low Back Pain
Keywords: low back pain; pediatric; gymnasts
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Female gymnasts with low back pain: Subset of competitive female gymnasts who report significant low back pain that affects their ability to perform gymnastics.
- Female gymnasts without low back pain: Subset of competitive female gymnasts who deny significant low back pain that affects their ability to perform gymnastics.

SUMMARY:
Low back pain is a common condition in children who perform gymnastics. Commonly, the injury is not the result of a specific injury, but is a stress injury to the lumbar spine. Regional interdependence is a theory that suggests when adjacent joints and muscles are not working properly increased stress is placed on a particular joint. This theory would suggest that if a patient did not have enough hip extension to perform a back bend increased motion would occur in the lumbar spine allowing the gymnast to complete the technique. Currently, no research links impairments in other joints to low back pain in gymnasts.

This is a cross sectional study assessing the relationship between gymnast with back pain and flexibility and strength of the shoulder and hip joints. Investigators will travel to a local gymnastics training centers and assess the gymnasts' strength and flexibility of the the hips and shoulders. The gymnast will also fill our a questionnaire assessing if they have had back pain in the past month and how much has it limited their ability to participate in gymnastics. Investigators will be blinded to the results of this survey.

The goal of this research study is to see if there are any link between strength and flexibility of the hips, and shoulders and gymnasts with low back pain. The investigators hypothesize that gymnasts who demonstrates impairments in strength and flexibility of the hips, or shoulders will be more likely to have complaints of low back pain.

DETAILED DESCRIPTION:
Female gymnasts will fill out a survey prior having their strength and flexibility tested. The investigators will be blinded to the results of the survey.

The questionaire asked the gymnasts several questions:

1. Age
2. Years in Gymnastics
3. At what level did you last compete?
4. On average how many hours per week do you participate in gymnastics?
5. Have you had any back pain in the past month that has affected your ability to participate in gymnastics?
6. If you answered yes to the last question: please rate your ability to participate in gymnastics with back pain?(0 represents unable to perform gymnastics and 100 represents no difficulty participating in gymnastics

After the gymnast complete the survey the investigators will assess the flexibility and strength of their shoulder and hip muscles. Investigators will be blinded to survey results. Evaluation measures will be performed in a randomized manner. Subjects will randomly perform shoulder or hip testing first (determined by flip of coin). Flexibility and strength testing will also be determined randomly (determined by flip of coin).

Evaluation measures

Shoulder Flexibility Passive Motion test:

* Prior to shoulder flexibility testing, the gymnast's arm length is measured from the tip of the acromion process to a ½ inch wooden dowel grasped by both hands while holding their shoulders flexed to 90 degrees.
* For testing, the gymnast lies prone on a firm floor with their chin and nose touching the floor.
* Both arms are held parallel to the body with the shoulders flexed to 180 degrees.
* The gymnast grasps the ½ inch dowel with and overhand grip and the tips of her thumbs are touching.
* The evaluator maximally flexes the gymnasts shoulders while maintaining wrist in neutral position, elbows extended and their nose and chin in contact with the floor.
* Once the gymnast's arms are raised to maximum height, the distance from the dowel, where the thumbs are touching, to the floor is measured and recorded to the nearest ½ centimeter using a rigid measuring stick.
* The Shoulder flexibility Passive Motion test raw score is calculated my dividing the dowel height attained by the length of the gymnast's arm.

Shoulder Flexibility Active Motion test:

* Prior to shoulder flexibility testing, the gymnast's arm length is measured from the tip of the acromion process to a ½ inch wooden dowel grasped by both hands while holding their shoulders flexed to 90 degrees.
* For testing, the gymnast lies prone on a firm floor with their chin and nose touching the floor.
* Both arms are held parallel to the body with the shoulders flexed to 180 degrees.
* The gymnast grasps the ½ inch dowel with and overhand grip and the tips of her thumbs are touching.
* The gymnast is asked to maximally flex their shoulders while maintaining wrist in neutral position, elbows extended and their nose and chin in contact with the floor.
* Once the gymnast has raised their arms to the maximum height, the distance from the dowel, where the thumbs are touching, to the floor is measured and recorded to the nearest ½ centimeter using a rigid measuring stick.
* The Shoulder flexibility test raw score is calculated my dividing the dowel height attained by the length of the gymnast's arm.

Hip Extension Flexibility test (Thomas test):

* Prior to hip extension flexibility testing, the gymnast lays flat on the examination table with legs extended. The examiner places the digital inclinometer on the anterior portion of the mid-thigh and zeros the inclinometer. The examiner marks the gymnast's skin at the distal most portion of the inclinometer in contact with the gymnast.
* Hip extension flexibility will be measured by using the modified Thomas test.
* The gymnast is instructed to sit as close to the edge of the examination table as possible.
* The gymnast supports their contralateral thigh with their arms and, with the assistance of the examiner, slowly rolls backward onto the table.
* The contralateral hip is flexed to the point that the gymnast's lumbar lordosis is flattened, and the right limb is allowed to hang unsupported off the table.
* The examiner palpates the lumbar spine to confirm that it remains in contact with the table.
* Thigh position is also monitored to prevent abduction of the thigh.
* When the final test position is achieved the examiner places the inclinometer on the gymnast's anterior thigh in line made prior to testing.
* 0 degrees indicates the gymnast's thigh is parallel to the horizon. If the thigh was above horizontal the number from the digital inclinometer will be read as negative. If the thigh is below horizontal the number will be positive.

Dynamometer Testing:

After having received standardized instructions, subjects will perform a series of familiarization trials consisting of three submaximal contractions per side. Then maximal voluntary contraction strength will be measured. The side tested first will be randomized within each test session. All maximal voluntary contraction strength data provided by the dynamometer (in kilograms) will be normalized to body weight.

Shoulder Flexion Strength test:

* Strength testing will be performed with hand held dynamometer stabilized by the examiner.
* For testing, the gymnast lies prone on a firm floor with their chin and nose touching the floor.
* Both arms are held parallel to the body with the shoulders flexed to 180 degrees.
* The gymnast grasps the ½ inch dowel with and overhand grip and the tips of her thumbs are touching.
* The dynamometer pad will be will located on the ½ inch dowel where the gymnasts thumbs meet.
* The gymnast is asked to maximally flex their shoulders pressing the dowel into the dynamometer pad as hard as they can while maintaining wrist in neutral position, elbows extended and their nose and chin in contact with the floor.
* Two to three maximal voluntary contraction trials will be permitted. A third trial is completed only if the difference between the first two maximal voluntary contractions is >10%.
* The duration of these contractions will be 5 seconds, and thirty seconds of rest will be given between trials.
* If gymnast is unable to actively flex shoulders to 180 degrees the strength test will be scored as 0.

Isometric maximal voluntary contraction strength of the hip muscles will be measured with a portable dynamometer fixed to a custom made frame. The custom-made frame is firmly fixed to a physical therapy treatment table with use of screw clamps. The frame consisted of two vertical bars and 1 horizontal bar attached to the vertical bars so as to be perpendicular to the extremities. The dynamometer is fixed to the horizontal bar so as the testing pad can be positioned properly for testing.

.

Hip Extension Strength Dynamometer Test:

* Gymnast is in prone position on examination table with tested leg knee fully extended. Tested hip is in 5 degrees of extension with the knee in full extension.
* The dynamometer is fixed using the custom made frame
* The center of the dynamometer pad will be on the posterior aspect of the calcaneus
* Gymnast is told to stabilize themselves by holding onto the examination table
* Gymnasts is instructed to push as hard as they can against the dynamometer testing pad.
* Two to three maximal voluntary contraction trials will be permitted. A third trial is completed only if the difference between the first two maximal voluntary contractions is >10%.
* The duration of these contractions will be 5 seconds, and thirty seconds of rest will be given between trials.

Hip Abduction Strength Dynamometer test:

* Gymnast is in sidelying position on examination table with tested leg knee fully extended.
* The contralateral hip and knee joints will be positioned at approximately 30 degrees of flexion for stability and comfort.
* Tested hip is in 10 degrees of abduction with the knee in full extension.

  •. The center of the dynamometer pad will be located 5 cm proximal to the lateral femoral condyle.
* Gymnast is told to stabilize themselves by holding onto the examination table.
* Gymnast is instructed to push as hard as they can against the dynamometer testing pad.
* The examiner will inspect the whole body position during the maximal voluntary contraction trials to ensure minimal compensation from pelvic rotation and flexion and rotation about the hip. If the examiner judges too much compensation, that test will not be recorded and the subject will be reinstructed in proper testing form.
* Two to three maximal voluntary contraction trials will be permitted. A third trial is completed only if the difference between the first two maximal voluntary contractions is >10%.
* The duration of these contractions will be 5 seconds, and thirty seconds of rest will be given between trials.

ELIGIBILITY:
Inclusion Criteria:

* At least 7 years old
* Level 5 or higher gymnast
* Female

Exclusion Criteria:

* Patient with a injury to the shoulder, or hips that prevents them from performing gymnastics.
* Patients who are unable to follow directions.

Min Age: 7 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Competitive female gymnasts. Females who perform gymnastics at local gymnastics training centers.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Presence of low back pain in past month | Baseline
  Presence of significant low back pain that has affected gymnastics ability at time of evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell C Selhorst, DPT, Principal Investigator — Nationwide Childrens Hospital
Locations (1):
- Buckeye Gymnastics, Powell, Ohio, United States

REFERENCES:
- [Background] Thorborg K, Petersen J, Magnusson SP, Holmich P. Clinical assessment of hip strength using a hand-held dynamometer is reliable. Scand J Med Sci Sports. 2010 Jun;20(3):493-501. doi: 10.1111/j.1600-0838.2009.00958.x. Epub 2009 Jun 23. PMID 19558384
- [Background] Sleeper MD, Kenyon LK, Casey E. Measuring fitness in female gymnasts: the gymnastics functional measurement tool. Int J Sports Phys Ther. 2012 Apr;7(2):124-38. PMID 22530187
- [Background] Widler KS, Glatthorn JF, Bizzini M, Impellizzeri FM, Munzinger U, Leunig M, Maffiuletti NA. Assessment of hip abductor muscle strength. A validity and reliability study. J Bone Joint Surg Am. 2009 Nov;91(11):2666-72. doi: 10.2106/JBJS.H.01119. PMID 19884441